CLINICAL TRIAL: NCT01034748
Title: A Phase One Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism And Excretion Of [14C]PF-00299804 in Healthy Male Volunteers
Brief Title: A Radiolabeled Mass Balance Study Of [14C]PF-00299804 In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A7471020
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Radiolabelled; Mass Balance; Healthy Volunteers; Pharmacokinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single 45 mg oral dose of [14C]PF-00299804
  Interventions: Drug: [14C]PF00299804

INTERVENTIONS:
Drug: [14C]PF00299804 — Single 45 mg oral dose of radiolabelled PF-00299804

SUMMARY:
This is single dose study of radiolabeled [14C]PF-00299804 in healthy male volunteers to study the absorption, distribution, metabolism and elimination of PF-00299804.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.)
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products within 3 months of screening or a positive urine cotinine test at Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* 12 lead ECG demonstrating QTc >450 msec at Screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Subjects enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry.
* Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subject is the investigator or a sub investigator, research assistant, pharmacist, study coordinator, other staff, or a relative of study personnel directly involved with the conduct of the study.
* Subjects who are believed to be unable and/or unlikely to comprehend and follow the trial protocol.
* Subjects with a history of irregular bowel movements eg, regular episodes of diarrhea or constipation, irritable bowel syndrome (IBS) or lactose intolerance.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: Estimation of PK parameters (Cmax, Tmax, AUClast, AUCinf, t1/2, CL/F and Vd/F, as data permit) for PF 00299804, major metabolites (if possible), and total radioactivity. | 1 month
Mass balance: Calculation of % total recovery of total radioactivity in urine and feces; calculation of % dose excreted of major metabolites (if possible). | 1 month
Metabolic profiling / metabolite identification: Metabolic profile of PF 00299804 derived from plasma, urine and fecal samples; identification of major metabolites of PF-00299804 in plasma, urine and/or feces if possible. | 1 month

SECONDARY OUTCOMES:
Safety laboratory tests, physical examination, vital signs, ECGs, concomitant medications and adverse event monitoring. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471020&StudyName=A%20Radiolabeled%20Mass%20Balance%20Study%20Of%20%5B14C%5DPF-00299804%20In%20Healthy%20Male%20Volunteers